CLINICAL TRIAL: NCT04944615
Title: IVUS-CTO: Comparison of the Effect of Intravascular Ultrasound-guided Versus Angiographic-guided Drug-eluting Stent Implantation on Long-term Clinical Outcomes in Patients With Chronic Complete Occlusion of Coronary Artery Disease: a Prospective, Multicenter, Randomized Controlled Clinical Study
Brief Title: To Evaluate Whether IVUS-guided Drug-eluting Stent (DES) Implantation Leads to Better Clinical Outcomes Compared to Conventional Angiography in the Treatment of Chronic Complete Occlusion (CTO) Disease.
Acronym: CRUISE-CTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CCRF Inc., Beijing, China (Industry)
Collaborators: BSC International Medical Trading (Shanghai) Co., Ltd. (Other)
Responsible Party: Principal Investigator, Yaling Han, M.d., Ph.D., Academician/chief physician, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Record Dates: First submitted 2021-06-01; First posted 2021-06-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Chronic Total Occlusion of Coronary Artery
Keywords: TIMI flow = grade 0 coronary artery disease with a duration greater than 3 months.

STUDY DESIGN:
Intervention Model Description: Patients were enrolled when the guide wire successfully passed through the CTO lesion (defined as: the guide wire successfully passed through the CTO lesion and reached the distal true lumen as confirmed by angiography).
  Once patients have signed the informed consent form and met all clinical and angiographic inclusion criteria and did not meet all clinical and angiographic exclusion criteria, and the guide wire has successfully passed the CTO lesion, they may be considered for participation in the study and randomized.
  The random grouping arrangement is computer generated using a quasi-random number generator.
  All randomized subjects will be assigned a unique identification number. Randomized replacement blocks will be used to ensure that the distribution of treatment within each layer is approximately balanced.
  The study also used the Interactive Voice Response System (IVRS)/Interactive Internet Response System (IWRS) to assign subjects to the study device treatment group.
Masking Description: During the study, it is difficult for researchers, operators and patients to blind the method due to objective reasons.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravascular ultrasound guidance (Experimental): All targeted CTO lesions will be examined and documented using a commercially available IVUS catheter (Opticross HD) according to its instructions (if not contraindicated, preoperative vasodilation with nitroglycerin to prevent spasm).
  IVUS examination must be performed at least once before and after stent implantation.
  Interventions: Procedure: The guidewire successfully passed the CTO lesion
- Angiographic guidance (Active Comparator): The patient will choose the appropriate length and diameter of the stent to be implanted by visual estimation. All commercially available drug-eluting stents (except first-generation DES, such as Taxus, Excel, Partner, Firebird, etc.) can be used. DES with high quality clinical evidence is strongly recommended. The type, diameter, and length of the stent are determined by the surgeon. The stent length should be selected to ensure complete coverage of the CTO lesion. If dissection is present, additional stents are implanted. Repeat angiograms were performed immediately after surgery in the same view as before surgery.
  Interventions: Procedure: The guidewire successfully passed the CTO lesion

INTERVENTIONS:
Procedure: The guidewire successfully passed the CTO lesion — The successful passage of the guide wire through the CTO lesion was defined as: the guide wire successfully passed through the CTO lesion and reached the distal true lumen as confirmed by angiography.
  Aspirin load dose (300 mg), clopidogrel load dose (300 mg), or ticagrelor load dose (180 mg) is recommended for all subjects prior to stent implantation and is recommended to be taken at least 6 hours prior to surgery.
  Other Names: Load dose administration

SUMMARY:
This study aims to evaluate the treatment of Chronic total occlusion (CTO) disease. Whether Intravascular Ultrasonography (IVUS) guiding the implantation of drug-eluting stents (DES) will provide better long-term clinical outcomes compared with conventional angiography

DETAILED DESCRIPTION:
The study was a prospective, multicenter, open-label, two-arm, 1:1 randomized controlled, well-designed clinical study.

According to the sample size calculation, a total of 1448 patients with primary CTO lesions were required to participate in the study after the guide wire successfully passed through the lesion (defined as: angiographic indication that the guide wire successfully passed through the CTO lesion and reached the distal true lumen).

The study will be conducted at no more than 45research centers. With competitive enrolment, a maximum of 500 patients can be enrolled at each center or until the study is completed, whichever comes first.

It is recommended that each center enroll at least 20 patients.

ELIGIBILITY:
Clinical inclusion criteria:

1. At least 18 years old
2. Subjects will understand the test requirements, treatment and surgery, and can provide written informed consent
3. Subjects with clinical symptoms of ischemic heart disease or evidence of myocardial ischemia associated with CTO target vessels and scheduled to undergo Percutaneous coronary intervention (PCI)
4. Subjects will receive percutaneous coronary intervention
5. Subjects are willing to accept all treatment and follow-up evaluations required by the protocol

Inclusion criteria for angiography:

1. Primary coronary artery CTO lesion with visible collateral circulation
2. Estimation of the time to complete occlusion (TIMI grade 0) ≥3 months based on clinical history and/or comparison with historical angiography or ECG
3. It is suitable for target lesions of 2.25-4.0mm stent implantation
4. The length of CTO lesion should be greater than 20mm

Clinical exclusion criteria:

1. Pregnant and lactating women
2. Severe coronary artery disease, not suitable for PCI
3. Patients with acute myocardial infarction less than 7 days
4. Long-term contraindications to DAPT (at least 1 year)
5. Known renal insufficiency.20 mL/min / 1.73 ㎡)
6. Left ventricular ejection fraction <35% or cardiogenic shock
7. The ICD implanted/CRT
8. Severe bleeding or stroke within 6 months
9. Have a history of allergy to iodine contrast agents or any known allergy to clopidogrel, ticagrelor, aspirin, or heparin
10. Subjects have been diagnosed or suspected of liver disease, including laboratory evidence of hepatitis
11. Valvular heart disease significantly affecting hemodynamics, hypertrophic cardiomyopathy, restrictive cardiomyopathy, or congenital heart disease
12. Diseases that researchers believe may seriously harm patients, such as cancer and mental illness;Or the patient's life expectancy is less than one year and the follow-up cannot be completed;Or other conditions that researchers think might have confounded the results
13. Participate in any other ongoing trial or intend to participate in another clinical trial of a drug or device within 12 months after baseline surgery

Angiographic exclusion criteria:

1. The target lesion is located in the left main artery
2. No visible collateral circulation in CTO lesions
3. Target lesion is venous or arterial bypass graft
4. The target vessel occlusion time (TIMI grade 0) < 3 months can be determined

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1448 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2031-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | The study design was event-driven. When a predetermined number of primary endpoints (number of MACE events = 291) occurs (expected 3 years), the study termination procedure will be initiated and this data will be used for primary end point analysis.
  All causes of death, myocardial infarction, stent thrombosis (ARC clear/probable), and clinically driven target vessel revascularization

SECONDARY OUTCOMES:
Cardiogenic death | 30 days, 6 months, 12 months, 24 months, 36 months, 48 months after surgery
  This includes acute myocardial infarction, cardiac perforation/tamponade, arrhythmia or conduction abnormalities, cerebrovascular accidents at discharge or suspected operating-related cerebrovascular accidents, death from surgical complications, including hemorrhage, vascular repair, transfusion reaction, or bypass surgery, or any death of cardiac origin that cannot be ruled out.
Nonfatal myocardial infarction | 30 days, 6 months, 12 months, 24 months, 36 months, 48 months after surgery
  Nonfatal myocardial infarction
Target lesion revascularization | 30 days, 6 months, 12 months, 24 months, 36 months, 48 months after surgery
  Target lesion revascularization is any ischemia-driven repetitive percutaneous coronary intervention to improve blood flow to a successfully treated target lesion or to bypass the target vessel and use a graft distally to the successfully treated target lesion.
  If the target lesion diameter is ≥50% stenosis as assessed by QCA and there is clinical or functional ischemia that cannot be explained by other coronary or graft lesions, vascularization will be considered to be induced by ischemia.
Target vessel revascularization | 30 days, 6 months, 12 months, 24 months, 36 months, 48 months after surgery
  Target vessel revascularization is defined as repeated intervention in the vessel where the target lesion is located in reference to target lesion revascularization
Target lesion failure | 30 days, 6 months, 12 months, 24 months, 36 months, 48 months after surgery
  Target lesion failure refers to target lesion revascularization, target vascular-related MI (Q wave and non-Q wave) or (cardiac) death due to ischemia
Target vessel failure | 30 days, 6 months, 12 months, 24 months, 36 months, 48 months after surgery
  Target vessel failure refers to target vessel revascularization, target-related MI (Q wave and non-Q wave), or target-related (cardiac) death resulting from ischemia
Left ventricular function improved | Baseline period and one-year follow-up period
  Left ventricular ejection fraction at 1 year and changes from baseline to 1 year
Percentage stenosis of segmental and stent diameter | The follow-up period was 12 months
  Anangiographic percentage of insegment and instent diameter stenosis measured by QCA at 12 months postoperatively
Lumens in segmental vessels and stents were lost | The follow-up period was 12 months
  12 months postoperatively, angiographic measurements of intrasegmental and in-stent lumens by QCA were lost
Binary restenosis rate in segment and stent | The follow-up period was 12 months
  Binary restenosis refers to the previously treated stenosis diameter at the lesion site > 50%, including the original treatment area and proximal and distal areas adjacent to the QCA analysis segment
Minimum lumen diameters in segments and stents | The follow-up period was 12 months
  Minimum lumen diameters in segmental vessels and stents as measured by QCA 12 months postoperatively
QCA measurements were obtained immediately in the lumen | Baseline operative period
  Immediate luminal measurements of QCA during surgery were obtained
MLD measured by QCA | Baseline operative period
  MLD measured by QCA during surgery
Clinical success rate | Baseline operative period
  Clinical success was defined by visual evaluation of mean lesion diameter stenosis by the physician on 2 near-orthogonal projection angiography with TIMI blood flow grade 3.
  No nosocomial myocardial infarction, TVR or cardiac death occurred in 30% of patients

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Shenyang Military Region, Beijing, China